CLINICAL TRIAL: NCT04129372
Title: Evaluating "New Foods Take Time", a Classroom-based Curriculum Designed to Promote Tasting and Liking of Fruits and Vegetables Among Head Start Preschool Children
Brief Title: New Foods Take Time, a Curriculum Designed to Promote Tasting and Liking of Fruits and Vegetables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jennifer Savage Williams, Associate Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013066
Record Dates: First submitted 2019-10-09; First posted 2019-10-16 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Eating Behavior
Keywords: fruits; vegetables; food neophobia; preschool; children
MeSH Terms: conditions — Feeding Behavior; Avoidant Restrictive Food Intake Disorder

STUDY DESIGN:
Intervention Model Description: Classrooms will receive "New Foods Take Time", a series of 5 interactive lessons. Children, parents, and teachers will participate in the research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New Foods Take Time (Experimental): Head Start classrooms will receive "New Foods Take Time", a series of five interactive weekly lessons designed to promote children's willingness to try new foods, particularly fruits and vegetables. Lessons will be delivered by nutrition educations. Children will also receive three tastings per week of the new foods discussed during the lessons.
  Interventions: Behavioral: New Foods Take Time

INTERVENTIONS:
Behavioral: New Foods Take Time — New Foods Take Time is a series of 5 classroom lessons focused on increasing children's willingness to try fruits and vegetables.

SUMMARY:
The overall objective of this project is to conduct a preliminary evaluation of the "New Foods Take Time" Intervention in Head Start preschool classrooms.

DETAILED DESCRIPTION:
The overall objective of this project is to conduct a preliminary evaluation of the "New Foods Take Time" Intervention. This curriculum is designed to increase children's preference for and consumption of fruits and vegetables (FV) by encouraging children to try new FV and repeatedly taste these foods.

ELIGIBILITY:
Child Inclusion Criteria:

* Enrolled in a Head Start preschool center
* Between the ages of 2 and 5 years old

Child Exclusion Criteria:

* Food allergy or restriction to foods in the tastings

Parent Inclusion Criteria:

* Parent or primary caregiver of a child enrolled in the study
* Age 18 years or older
* English speaking

Parent Exclusion Criteria:

* None

Teacher Inclusion Criteria:

* Actively employed as an early childhood education provider in the Head Start classroom where the intervention is delivered
* Age 18 years or older

Teacher Exclusion Criteria:

* None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Change in number of foods tasted | Pre intervention and at conclusion of 5 week intervention
  Children will be presented with small portions of familiar and novel fruits and vegetables and be asked if they would like to taste them
Change in liking of study foods | Pre intervention and at conclusion of 5 week intervention
  For foods that children agree to taste, they will be asked to rate their liking of them on a three point likert-type scale ("Yummy", "Just ok", or "Yucky")
Change in self-competence to try new foods | Pre intervention and at conclusion of 5 week intervention
  Children will be presented with a series pairs of drawings with descriptions (e.g., "This boy likes to try new foods" and "This boy does not like to try new foods") and asked to select which is most like them.
Teacher acceptability of intervention | At conclusion of 5 week intervention
  Teachers will complete a questionnaire with scaled and open-ended questions about the feasibility and acceptability of the intervention

OTHER OUTCOMES:
Child body mass index | Measured once at any time between enrollment and conclusion of 5 week intervention
  Height and weight will be measured and used to calculate body mass index (BMI). Age and sex specific percentiles/z-scores will be calculated using CDC growth standards.
Parent report of child neophobia | Measured once at any time between enrollment and conclusion of 5 week intervention
  Parents will complete a survey about their child's eating behavior
Parent report of food insecurity | Measured once at any time between enrollment and conclusion of 5 week intervention
  Parents will complete the USDA food security questionnaire
Change in intake of study foods | Pre intervention and at conclusion of 5 week intervention
  The number of pieces of each food eaten during the tasting procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Savage, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available from the principal investigator upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication of primary outcomes
Access Criteria: Requests for access to the data will be reviewed and approved at the principal investigator's discretion.